CLINICAL TRIAL: NCT04772508
Title: Efficacy of Subgingivally Placed Amnion Membrane With and Without Taurine as an Adjunct to Scaling and Root Planing in the Treatment of Chronic Periodontitis
Brief Title: Effect of Amnion Membrane With and Without Taurine on GCF TNF α Level.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DR SURINDER SACHDEVA, PROFESSOR, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13/395
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Periodontitis
Keywords: periodontitis; taurine; amnion membrane
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; Taurine

STUDY DESIGN:
Intervention Model Description: Group A (Control): 15 sites received only SRP, Group B: 15 sites received SRP with subgingival placement of amnion membrane, Group C: 15 sites received SRP with subgingival placement of Amnion membrane hydrated with Taurine.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and statistician are masked about treatment modality
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Sham Comparator): 15 sites received only scaling and root planing
  Interventions: Procedure: Scaling and root planing
- Group B (Active Comparator): 15 sites received scaling and root planing with subgingival placement of amnion membrane
  Interventions: Procedure: Scaling and root planing; Biological: Amnion membrane
- Group C (Active Comparator): 15 sites received scaling and root planing with subgingival placement of amnion membrane hydrated with Taurine
  Interventions: Procedure: Scaling and root planing; Biological: Amnion membrane; Drug: Taurine

INTERVENTIONS:
Procedure: Scaling and root planing — 15 sites with periodontal pockets ≥ 5mm received only SRP
  Other Names: SRP
Biological: Amnion membrane — 15 sites with periodontal pockets ≥ 5mm received SRP along with placement of amnion membrane.
  Other Names: AM
  Arms: Group B; Group C
Drug: Taurine — 15 sites with periodontal pockets ≥ 5mm received SRP along with placement of amnion membrane hydrated with taurine.
  Other Names: T
  Arms: Group C

SUMMARY:
45 sites in 15 patients with periodontal pockets ≥ 5mm were selected. These selected sites were divided into 3 groups as Group A, B and C.

DETAILED DESCRIPTION:
Group A (Control): 15 sites received only SRP, Group B: 15 sites received SRP with subgingival placement of amnion membrane, Group C: 15 sites received SRP with subgingival placement of Amnion membrane hydrated with Taurine.

ELIGIBILITY:
Inclusion Criteria:

•Systemically healthy patients with sites showing probing depth (PD) ≥ 5mm, clinical attachment level (CAL) ≥ 4 mm, and vertical bone loss ≥ 3 mm on intraoral periapical radiographs with no history of periodontal therapy or use of antibiotics in the preceding 6 months

Exclusion Criteria:

* Any systemic disease that could influence the outcome of periodontal therapy.
* Smokers, alcoholics & patients with other adverse habits.
* Pregnant or nursing women.
* Any known allergy or hypersensitivity to any product used in the study.
* Patients on long term systemic therapy (antibiotics, anti-inflammatory and any other).

Ages: 29 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
TNF-α level | changes from baseline to 45 days
  TNF-α level in Gingival crevicular fluid
Probing pocket depth (PPD) | changes from baseline to 45 days
  Probing pocket depth at selected site
Relative attachment level (RAL) | changes from baseline to 45 days
  Relative attachment level from stent to base of the pocket

SECONDARY OUTCOMES:
Plaque index (PI) | changes from baseline to 45 days
  Plaque index (PI) - Silness and Loe 1964 site specific
Gingival index (GI) | changes from baseline to 45 days
  Gingival index (GI) - Loe and Silness 1963 site specific
Bleeding on probing (BOP) | changes from baseline to 45 days
  Bleeding on probing (BOP): Muhlemann HR & Son 1971 sit specific

CONTACTS AND LOCATIONS:
Overall Officials: surinder sachdeva, M.D.S., Study Director — PROFESSOR
Locations (1):
- Department of Periodontology, M.M. College of Dental Sciences and Research., Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giris M, Depboylu B, Dogru-Abbasoglu S, Erbil Y, Olgac V, Alis H, Aykac-Toker G, Uysal M. Effect of taurine on oxidative stress and apoptosis-related protein expression in trinitrobenzene sulphonic acid-induced colitis. Clin Exp Immunol. 2008 Apr;152(1):102-10. doi: 10.1111/j.1365-2249.2008.03599.x. Epub 2008 Jan 28. PMID 18241224
- [Background] Gultekin SE, Senguven B, Sofuoglu A, Taner L, Koch M. Effect of the topical use of the antioxidant taurine on the two basement membrane proteins of regenerating oral gingival epithelium. J Periodontol. 2012 Jan;83(1):127-34. doi: 10.1902/jop.2011.100568. Epub 2011 May 16. PMID 21574832